CLINICAL TRIAL: NCT00271115
Title: The Effect of Kangaroo Holding on Maternal Stress Levels
Brief Title: Kangaroo Holding and Maternal Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 25165
Record Dates: First submitted 2005-12-21; First posted 2005-12-30 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Premature Birth; Maternal Stress
Keywords: Kangaroo holding; Kangaroo care; Maternal stress levels; Premature birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moms w/preterm infants (Other): Mothers of preterm infants who are admitted to the newborn intensive care unit.
  Interventions: Behavioral: Kangaroo Holding

INTERVENTIONS:
Behavioral: Kangaroo Holding — Mothers will be asked to Kangaroo hold their infants two times during the first week of life.

SUMMARY:
The primary objective is to determine if kangaroo holding in the first week after birth influences the stress levels of mothers who have delivered their infants prematurely and who require admission to the Special Care Nursery (SCN).

Hypothesis: There will be a decrease in maternal stress levels as perceived by mothers and as reflected in their blood pressures and heart rates after kangaroo holding their premature infants in the SCN.

DETAILED DESCRIPTION:
This study builds on known observations by previous researchers that the birth and hospitalization of premature infants creates stressful events in the lives of parents (Shields-Poe & Pinelli, 1997). The challenge for health care workers is to provide for the physical and psychological needs of infants within a highly technological setting such as the SCN. It is necessary to facilitate effective bonding between parents and infants. Effective bonding is linked with successful parenting role development. Stress can alter the development of a positive parental role.

Kangaroo holding, or skin-to-skin holding, involves placing a diaper clad infant vertical and prone between a mother's breasts (Affonso, 1993). As evidenced by the literature, stress can have an altering effect on the maternal attachment role psychologically and place physical demands on the cardiovascular system. Kangaroo care is one variable that may change the perception of maternal stress during preterm hospitalization by assisting mothers to gain control of the parental role, permitting maternal bonding and reducing maternal separation as well as potentially decreasing the allostatic load as associated with physiologic stress.

This study will compare maternal perceived stress levels before and after kangaroo holding during the first week of life. Mothers who are enrolled in this study will be asked to Kangaroo hold their infants at least two times during the first week of life. The first kangaroo hold will take place with the first 48 hours of life. The second kangaroo hold will take place between day of life five and seven. Mothers may kangaroo hold their infants more than two times, however this study will only examine the kangaroo holding sessions that take place at the two times specified above. This study includes both physiologic and psychologic measurements. Mothers will have their blood pressure and heart rate measured before and after each of the two kangaroo holding sessions. These mothers will also be asked to complete a self-report stress inventory scale prior to the first kangaroo holding session (first 48 hours of infant's life) and again after the second kangaroo holding session (infant's day of life five to seven).

ELIGIBILITY:
Inclusion Criteria:

Mothers:

* Delivered a premature infant between 30 0/7 and 33 6/7 weeks gestation
* 20 to 40 years old
* English speaking

Infants:

* Admitted to Special Care Nursery and on a monitor
* Medically stable enough to be held (determined by health care team)

Exclusion Criteria:

Mothers:

* Multiple birth
* Eclampsia
* Pre-existing hypertension or at risk (BP above 140/90)
* Pre-existing cardiac disease
* HELLP syndrome, or uncontrolled medical condition during pregnancy
* Use of magnesium sulfate for blood pressure control prior to delivery
* Known depression or treatment with antidepressants

Infants:

* Congenital anomalies
* Use of NCPAP or mechanical ventilation
* medically unstable (as determined by health care team)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-09; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change in perceived maternal stress after kangaroo holding. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Karen A. Hall, BSN, RNC, Principal Investigator — Christiana Care Health Systems
Locations (1):
- Christiana Hospital - Special Care Nursery, Newark, Delaware, United States

REFERENCES:
- [Background] Affonso D, Bosque E, Wahlberg V, Brady JP. Reconciliation and healing for mothers through skin-to-skin contact provided in an American tertiary level intensive care nursery. Neonatal Netw. 1993 Apr;12(3):25-32. PMID 8474409
- [Background] Miles MS, Funk SG, Carlson J. Parental Stressor Scale: neonatal intensive care unit. Nurs Res. 1993 May-Jun;42(3):148-52. PMID 8506163
- [Background] Miles MS, Funk SG, Kasper MA. The stress response of mothers and fathers of preterm infants. Res Nurs Health. 1992 Aug;15(4):261-9. doi: 10.1002/nur.4770150405. PMID 1496151